Title:

Status: Approved, Version: 1.0

Approved Date: 19 Nov 2020

## Statistical Analysis Plan for Protocol CLY935-E006 / NCT04631796

Protocol Title: Clinical Characterization of an Investigational Soft Silicone

Hydrogel Contact Lens

**Template Version:** Version 1.0

**Approvals:** See last page for electronic approvals

This is the original (Version 1.0) Statistical Analysis Plan for this study. This version of the Statistical Analysis Plan is based on Version 1.0 of the study protocol.

Document ID: V-CLN-0003152 Status: Approved, Version: 1.0 Approved Date: 19 Nov 2020

Page 2 of 13

#### **Executive Summary:**

Key Objectives:

The primary objective of this study is to evaluate the overall clinical performance of an investigational silicone hydrogel contact lens over 2 weeks of daily wear.

Decision Criteria for Study Success:

Decision criteria for study success are not applicable for this study.

Status: Approved, Version: 1.0 Approved Date: 19 Nov 2020

# **Table of Contents**

| Sta | atistical A | nalysis Plan for Protocol CLY935-E006 | 1 |
|---|---|---|---|
| Ta | ble of Co | ntents | 3 |
| Li | st of Table | es | |
| 1 | STUDY | OBJECTIVES AND DESIGN | 5 |
| | 1.1 | Study Objectives | |
| | 1.2 | Study Description | |
| | 1.3 | Randomization | |
| | 1.4 | Masking | |
| 2 | ANALY | SIS SETS | 6 |
| | 2.1 | Safety Analysis Set | 6 |
| 3 | SUBJEC | CT CHARACTERISTICS AND STUDY CONDUCT SUMMARIES | |
| 4 | EFFICACY ANALYSIS STRATEGY | | |
| | 4.1 | | |
| | 4.2 | Effectiveness Hypotheses | |
| | 4.3 | Statistical Methods for Effectiveness Analyses | |
| | | 4.3.1 Primary Effectiveness Analyses | |
| 5 | SAFET | ETY ANALYSIS STRATEGY9 | |
| | 5.1 | Safety Endpoints | |
| | 5.2 | Safety Hypotheses10 | |
| | 5.3 | , and the second se | |
| | | 5.3.1 Adverse Events | |
| | | 5.3.2 Biomicroscopy Findings/Slit Lamp Examination | |
| | | 5.5.5 Device Deficiencies | 11 |
| 8 | REFERI | ENCES | 11 |
| 0 | | | |

| V-CLN-000 | | Approved Date: 19 Nov 2020 | Page 4 of 13 |
|---|---|---|---|
| 9 REVISI | ON HISTORY | | 11 |
| 10 APPEN | DIX | | 12 |
| | | List of Tables | |
| Table 1–1 | Study Description Su | mmary | 5 |
| Table 10-1 | Schedule of Study Pr | ocedures and Assessments | 12 |

Status: Approved, Version: 1.0 Approved Date: 19 Nov 2020

#### 1 STUDY OBJECTIVES AND DESIGN

## 1.1 Study Objectives

The primary objective of this study is to evaluate the overall clinical performance of an investigational silicone hydrogel contact lens over 2 weeks of daily wear.

## 1.2 Study Description

Key components of the study are summarized in Table 1-1.

Table 1–1 Study Description Summary

| Study Design | Prospective, single group, bilateral, open-label |
|---|---|
| Study Population | Volunteer subjects aged 18 or over who are habitual spherical weekly/monthly soft contact lens wearers, have at least 3 months of contact lens wearing experience, and who wear their habitual contact lenses at least 5 days per week and at least 8 hours per day. |
| | Target to complete: 30 Planned to enroll: ~36 |
| Number of Sites | ~3<br>US |
| Test Product | LID020098 |
| Control Product | None |
| Planned Duration of | Test Product: $\sim 14 \pm 2$ days |
| Exposure | |
| Visits | Visit 1 – Screening/Baseline/Order Spectacles |
| | Visit 2 Dispense Study Lens |
| | Visit 3 — Week 2 Follow-up/Exit |

1.3 Randomization

Randomization is not applicable for this study.

1.4 Masking

This is a single group, open-label study.

#### 2 ANALYSIS SETS

#### 2.1 Safety Analysis Set

Safety analyses will be conducted using the safety analysis set on a treatment-emergent basis. As such, the safety analysis set will include all subjects/eyes exposed to any study lenses evaluated in this study, except for the lenses used with the purpose of power optimization. For treatment-emergent safety analyses, subjects/eyes will be categorized under the actual study lenses exposed.

Status: Approved, Version: 1.0

Approved Date: 19 Nov 2020

Adverse events occurring from the time of informed consent but prior to first exposure to study lenses will be summarized in subject listings.

# 3 SUBJECT CHARACTERISTICS AND STUDY CONDUCT SUMMARIES

The following tables will be presented:

- Subject Disposition
- Analysis Set
- Subject Accounting
- Demographics Characteristics
- Baseline Characteristics (eg, lens brand, lens care brand)

4 EFFICACY ANALYSIS STRATEGY This study defines one primary endpoint . The Safety Analysis Set will be used for all effectiveness analyses. All data obtained in evaluable subjects/eyes will be included in the analysis. No imputation for missing values will be carried out. 4.1 Efficacy Endpoints **Primary Endpoint** The primary endpoint is front surface wettability, collected on a 5-point scale, for each eye.

Status: Approved, Version: 1.0

Approved Date: 19 Nov 2020



## 4.2 Effectiveness Hypotheses

#### **Primary Effectiveness**

No inferences are to be made on the primary effectiveness endpoint; therefore, no hypotheses are formulated.



## 4.3 Statistical Methods for Effectiveness Analyses

## 4.3.1 Primary Effectiveness Analyses

Descriptive statistics will be presented, to include frequencies and percentages in each grade as well for the combined category of Grade 0 and Grade 1.



Status: Approved, Version: 1.0

Approved Date: 19 Nov 2020

#### 5 SAFETY ANALYSIS STRATEGY

The focus of the safety analysis will be a comprehensive descriptive assessment of occurrence of adverse events as well as the other listed parameters. Therefore, no inferential testing will be done for the safety analysis.

## 5.1 Safety Endpoints

The safety endpoints are

- Adverse events (AE)
- Biomicroscopy Findings/Slit Lamp Examinations



• Device deficiencies

#### 5.2 Safety Hypotheses

There are no formal safety hypotheses in this study. The focus of the safety analysis will be a comprehensive descriptive assessment of safety endpoints listed in Section 5.1.

Status: Approved, Version: 1.0

Approved Date: 19 Nov 2020

## 5.3 Statistical Methods for Safety Analyses

The analysis set for all safety analyses is defined in Section 2.1.

#### **5.3.1** Adverse Events

The applicable definition of an AE is in the study protocol. All AEs occurring from when a subject signs informed consent to when a subject exits the study will be accounted for in the reporting.

Pre-treatment AEs will be separated from treatment-emergent AEs occurring during the study period. A pre-treatment AE is an event that occurs after signing informed consent but prior to exposure to study lenses. The period for treatment-emergent AE analysis starts from exposure to study lenses until the subject completes or is discontinued from the study.



## **5.3.2** Biomicroscopy Findings/Slit Lamp Examination

The following tables and supportive listings will be provided:

- Frequency and Percentage for Biomicroscopy Findings by Visit
- Incidence of Increased Severity by 2 or More Grades in Biomicroscopy Findings

- Listing of Subjects With Other Biomicroscopy Findings
- Listing of Subjects With Increased Severity by 1 Grade in Biomicroscopy Findings

Status: Approved, Version: 1.0

Approved Date: 19 Nov 2020

- Listing of Subjects With Increased Severity by 2 or More Grades in Biomicroscopy Findings
- Listing of Subjects with Infiltrates

#### **5.3.3** Device Deficiencies

The following tables and supportive listings will be provided:

- Frequency of Treatment-Emergent Device Deficiencies
- Listing of Treatment-Emergent Device Deficiencies
- Listing of Device Deficiencies Prior To Treatment Exposure



#### 8 REFERENCES

Not Applicable.

#### 9 REVISION HISTORY

This is the original (Version 1.0) Statistical Analysis Plan for this study. This version of the Statistical Analysis Plan is based on Version 1.0 of the study protocol.

## 10 APPENDIX

Table 10-1 Schedule of Study Procedures and Assessments

| Procedure/ Assessment | Visit 1<br>Screening/<br>Baseline/ | Visit 2 <sup>@</sup><br>Dispense | Visit 3 Week 2 Follow- up /Exit^ | USV |
|---|---|---|---|---|
| Informed Consent | X | | | |
| Demographics | X | | | |
| Medical History* | X | $X^{\infty}$ | X | X |
| Concomitant Medications* | X | $X^{\infty}$ | X | X |
| Inclusion/Exclusion | X | | | |
| Habitual lens<br>(brand, power*, lens care) | X | | | |
| Biomicroscopy | X | $X^{\infty}$ | X | X |
| Optimize study contact lens power | (X) | | | |
| Record study lens power | X | | | |
| Dispense study lenses* | | X | | (X) |
| | | • | • | - |

| Procedure/ Assessment | Visit 1<br>Screening/<br>Baseline/ | Visit 2 <sup>@</sup><br>Dispense | Visit 3<br>Week 2 Follow-<br>up /Exit^ | USV |
|---|---|---|---|---|
| Lens surface assessments (OD, OS): • Front surface wettability | | X | X | (X) |
| $\mathrm{AEs}^\Omega$ | X | X | X | X |
| Device deficiencies | X | X | X | X |
| Exit Form | (X) | (X) | X | (X) |



# Signature Page for V-CLN-0003152 v1.0



Signature Page for V-CLN-0003152 v1.0  $\,$